CLINICAL TRIAL: NCT05751551
Title: Feasibility and Effectiveness of a Personalized, Home-based Motor-cognitive Training Program in Community-dwelling Older Adults - a Pragmatic Pilot Randomized Controlled Trial
Brief Title: Feasibility and Effectiveness of a Home-based Motor-cognitive Training Program in Older Adults
Acronym: COCARE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swiss Federal Institute of Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BASEC-Nr. 2022-01746
Record Dates: First submitted 2022-12-01; First posted 2023-03-02 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: Aged; Independent Living
Keywords: Motor-cognitive intervention; Exergames; Telerehabilitation

STUDY DESIGN:
Intervention Model Description: This study will be conducted as an international, pragmatic pilot randomized controlled trial with two treatment arms, an intervention group (IG) and a control group (CG). It comprises a two-week intervention period in a rehabilitation clinic (for familiarization purpose) followed by a 10-week training period at home. It involves three trial partners: ETH Zürich, Don Carlo Gnocchi Foundation (Fondazione Don Carlo Gnocchi (FDG), Milan, Italy), and Materia Agecare ((MAT), Nicosia, Cyprus). The study conduction will take place at all three trial sites.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The intervention group will conduct a motor-cognitive training program added to usual care. The intervention starts with a familiarization period in rehabilitation centers (face-to-face supervision) for 2 weeks before participants of the intervention group continue it at home (under remote supervision) for 10 weeks with 3 training sessions per week for about 20-30 minutes.
  Besides, participants of the intervention group will participate in 3 assessment sessions: (1) T1 (baseline assessments), (2) T2 (pre-intervention, after familiarization period, before starting the home-based training), (3) T3 (post-intervention assessment).
  Interventions: Other: Personalized, home-based motor-cognitive training
- Control group (No Intervention): The control group will continue with their usual care. Apart from that, they will only attend 3 assessment sessions: (1) T1 (baseline assessments), (2) T2 (pre-intervention, after familiarization period, before starting the home-based training), (3) T3 (post-intervention assessment).

INTERVENTIONS:
Other: Personalized, home-based motor-cognitive training — The simultaneous motor-cognitive training in this study will be conducted in form of exergames (interactive video games) using Senso hardware (DIV-SENSO-H, Dividat GmbH, Schindellegi, Switzerland) - a stepping platform with 5 pressure sensitive plates which is connected to a screen. For the home-based training, a more mobile version of the Dividat Senso will be used: a foldable pressure-sensitive mat. In both devices, stimuli of exergames appear on the screen and the participants have to react by stepping in one of 4 directions (front, back, left, right).
  The motor-cognitive training approach allows targeting different cognitive functions such as attention, executive functions, memory, and visuo-spatial functions as well as balance, and strength.
  FITT-VP principles will serve as a guideline but based on the functional status of each participant (physical and cognitive), the training sessions will be personalized in terms of training content, intensity and duration.
  Arms: Intervention group

SUMMARY:
The goal of this clinical study is to test feasibility and effectiveness of a personalized, home-based motor-cognitive training program in community-dwelling older adults with prescription for rehabilitation.

Participants will conduct a motor-cognitive intervention program which is based on exergames (=interactive video games controlled by body movements), added to usual care for 2 weeks in rehabilitation centers (face-to-face supervision) and for 10 weeks at home (remotely supervised).

Researchers will compare an intervention group and a control group to compare possible effects of the home-based study intervention to the effect of usual care alone on cognition, physical functions, and balance confidence.

DETAILED DESCRIPTION:
Age-related declines in physical and cognitive functioning and the associated adverse outcomes such as restricted mobility, cognitive impairment, and falls ultimately result in a decrease of older adults' quality of life. In the light of the demographic change, these age-related declines gain special importance. Attempting to counteract these declines, previous studies have revealed that simultaneous motor and cognitive training may be equally or even more effective than separate training. In fact, simultaneous motor-cognitive training has shown to improve various physical, cognitive, and psychological functions in older adults - for instance balance, gait, executive control, processing speed, exercise enjoyment, depressive symptoms, and quality of life. However, most training programs are provided face-to-face, and accessibility is a major concern for older adults, especially in the post-pandemic era. Besides, due to the demographic change there is an increased need for long-term care/treatment challenging the health care system (in terms of finance, time, and personnel). Home-based rehabilitation programs offer a cost-effective solution to these problems.

However, previous research either investigated home-based training approaches based on separate motor-cognitive training, or, in case of simultaneous motor-cognitive training approaches, these have been tested in rather specific older populations (e.g., stroke survivors, Parkinson patients, older adults with cognitive impairment) or in healthy older adults. Yet, simultaneous motor-cognitive training in the home setting should be feasible and effective in a broader population of older adults especially in those without long-term access to traditional rehabilitation interventions accompanying them to full recovery. For this reason, this study aims to test the feasibility of a personalized, simultaneous motor-cognitive home-based training approach based on exergames for geriatric patients and to evaluate its effectiveness compared to usual care alone on physical and cognitive functions as well as on fall-related self-efficacy.

Potential participants will be screened and if eligible, asked if they are interested in partaking. All eligible and interested possible participants will be orally informed about the study and receive a written study information explaining the aim of the study, procedures, risks, and benefits of participation, as well as their rights and duties in case of participation. All participants will sign a written consent form, before any study-specific actions are performed.

The study will start with a baseline assessment. Then, participants will be randomized to either the intervention or the control group applying permuted block randomization. Subsequently, participants of the intervention group will perform 6 supervised, personalized motor-cognitive training sessions in a rehabilitation centre (ideally within 2 weeks) for about 20-30 minutes per session (familiarization period). Afterwards, participants of the intervention group will continue the training independently at home for 10 weeks, 3 times/week for about 20-30 minutes with the investigators supervising them via phone calls and regular personal visits. Physical and cognitive tests will be the basis for individual training plans which will further on be regularly adapted based on progression rules. All motor-cognitive training sessions in both intervention phases will be additional to usual care. The control group receives no additional training besides usual care. Participants of all groups will conduct 3 measurement sessions: (1) T1 (baseline assessments), (2) T2 (pre-intervention, after familiarization period, before starting the home-based training), (3) T3 (post-intervention assessment).

ELIGIBILITY:
Inclusion Criteria:

* Patient with prescription for rehabilitation (as in- or outpatient)
* Mini-Mental State Examination (MMSE) score ≥ 24
* Physically able to independently stand for at least 2 minutes
* Able to give informed consent as documented by signature
* Access to the internet at home
* Availability of a TV or large screen at home

Exclusion Criteria:

* Nursing home resident
* Mobility limitations or comorbidities impairing the ability to conduct a step-based motor-cognitive training
* Cognitive limitations or comorbidities impairing the ability to conduct a step-based motor-cognitive training
* Previous or current major psychiatric illness (e.g., schizophrenia, bipolar disorder, recur-rent major depression episodes)
* History of drug or alcohol abuse
* Terminal illness
* Severe sensory impairments
* Participation in another clinical trial/intervention study
* More than 2 weeks absence in the next 3-4 months

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2023-02-22 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-02-09 (Actual)

PRIMARY OUTCOMES:
Adherence rate | The adherence rate is assessed for all training sessions during the home-based intervention period, approximately for 10 weeks
  The duration of completed training sessions as percentages of the recommended duration of training sessions.
Attrition rate | The attrition rate is assessed during the data collection period, an average of 12 weeks
  Number of participants lost during the trial will be recorded (drop-outs in both groups)
Exergame Enjoyment Questionnaire (EEQ) | The EEQ is completed by the intervention group at T3 (post-measurement), thus about 12 weeks after study entry. The survey lasts 5-10 minutes
  The EEQ will be used to measure exergame enjoyment in participants of the intervention group. The questionnaire consists of 20 statements rated on a five-point Likert scale which results in a minimum possible score of 20 and a maximum possible score of 100. A higher score reflects greater exergame enjoyment.

SECONDARY OUTCOMES:
National Aeronautics and Space Administration-Task Load Index (NASA-TLX) | The NASA-TLX is completed by the intervention group at T3 (post-measurement), thus about 12 weeks after study entry. The survey lasts 5-10 minutes.
  The NASA-TLX is a self-report, multidimensional assessment tool that rates perceived workload in order to assess a task, a system, or other aspects of performance (in this case the DIVIDAT exergames). It contains five subscales: Mental Demand, Physical Demand, Temporal Demand, Performance, Effort and Frustration. Each subscale can be given a score between 0 and 20. A higher score reflects a higher workload.
Additional instructions | Additional instructions will be collected throughout the whole home-based intervention period, an average of 10 weeks
  It will be noted by the investigators whether additional instructions were required by the participants of the intervention group, meaning the instructions provided by the system were not enough.
Help requests | The number of help requests will be collected throughout the whole home-based intervention period, an average of 10 weeks
  The number of help requests by the participants of the intervention group will be noted by the investigators (e.g. in case of technical problems and understanding difficulties)
Intention to continue the training program | The assessment will take place at T3 (post-measurement), thus about 12 weeks after study entry. The survey takes about 30 seconds.
  The intention of participants of the intervention group to continue a similar home-based motor-cognitive training program after the project will be assessed with a single question. Answer will be given on a 5 point Likert scale (1=strongly disagree, 5=strongly agree)
Changes in psychomotor speed | The assessment takes place at T2 (pre-measurement) and T3 (post-measurement), thus about 2 and 12 weeks after study entry. The RTT lasts 5 minutes.
  The Reaction Time Test (RTT) conducted on the Dividat Senso measures psychomotor speed in terms of reaction to visual stimuli using the lower extremities in 6 directions (front right, front left, right, left, back right & back left). Reaction time is measured [ms].
Changes in selective attention | The assessment takes place at T2 (pre-measurement) and T3 (post-measurement), thus about after 2 and 12 weeks after study entry. The GoNogo Test lasts 5 minutes.
  To assess selective attention, the Go-Nogo Test will be conducted on the Dividat Senso. It evaluates the ability to suppress a response in the presence of irrelevant stimuli as well as the response latency during stimulus selection. Participants will be asked to react as fast as possible when a cross (x) is presented on the screen. However, in case the stimulus is a plus (+), they must remain still. Reaction time is measured [ms].
Changes in cognitive flexibility | The assessment takes place at T2 (pre-measurement) and T3 (post-measurement), thus about 2 and 12 weeks after study entry. The Flexibility Test lasts 5 minutes.
  Cognitive flexibility will be assessed with the Flexibility Test conducted on the Dividat Senso. The test assesses the flexibility of focused attention. Participants are instructed to react with a step towards a rounded figure and then an angular figure in an alternating manner. Reaction time is measured [ms].
Changes in static balance | The assessment takes place at T2 (pre-measurement) and T3 (post-measurement), thus about 2 and 12 weeks after study entry. The Sway Test lasts about 1-2 minutes.
  Static balance will be assessed with the Sway Test conducted on the Dividat Senso. Participants are instructed to stand as still as possible for 30 seconds. Movements of the COP are collected [in mm] - the shorter the better is the static balance.
Changes in dynamic balance | The assessment takes place at T2 (pre-measurement) and T3 (post-measurement), thus about 2 and 12 weeks after study entry. The Coordinated Stability Test lasts about 4 minutes.
  Dynamic balance will be assessed with the Coordinated Stability Test conducted on the Dividat Senso. At the beginning, participants are instructed to stand follow a shown figure with the COP. The trace length of the COP is recorded [in mm] - longer length means less dynamic balance.
Changes in functional balance | The assessment takes place at T2 (pre-measurement) and T3 (post-measurement), thus about 2 and 12 weeks after study entry. The TUG tests take about 2 minutes.
  To assess functional balance, the Timed up and go Test (TUG) will be performed. It requires the participant to rise from a standard arm chair, walk 3 meters at a comfortable walking speed, turn, return, and sit down on the chair again. Time to complete the task is recorded in seconds.
Changes in functional balance and dual task | The assessment takes place at T2 (pre-measurement) and T3 (post-measurement), thus about 2 and 12 weeks after study entry. The TUG-DT takes about 2 minutes.
  To measure dual task, the TUG dual task (TUG-DT) will be performed. Thereby, the motor task of the TUG test (getting up from a chair, walk three meters, come back and sit down again) will be complemented with a cognitive task. For the cognitive task, participants are instructed to count backwards from 90, subtracting 7 successively. The time until the patient is fully seated again is recorded. Then, the dual task cost will be calculated by determining the percentage at which the cognitive task interfered on the test performance (DTC [%] = 100*(simple task score - DT score)/simple task score).
Changes in strength (Lower limb power) | The assessment takes place at T2 (pre-measurement) and T3 (post-measurement), thus about 2 and 12 weeks after study entry. The STS tests takes about 2 minutes.
  Strength/Lower limb power will be assessed with the 30 seconds Sit-to-Stand Test (STS). The participants will start sitting on a chair and after a countdown, they must stand up straight and sit down again as many times as possible within a time frame of 30 seconds. Meanwhile, the number of times the patient fully stands up from the chair will be counted.
Changes in balance confidence | The assessment takes place at T2 (pre-measurement) and T3 (post-measurement), thus about 2 and 12 weeks after study entry. The survey lasts about 10 minutes.
  Balance confidence will be assessed with the Activities-specific Balance Confidence (ABC) Scale. The ABC Scale is measuring fall associated self-efficacy of a person in different activities and situations (e.g. stair climbing and walking on icy pavements).The scale is a 0% to 100% continuous response scale. The overall score is calculated by adding the item scores and dividing the total by 16 (i.e. the number of items). This total score ranges from 0% to 100% with.0% reflecting no confidence and 100% reflecting complete confidence.

CONTACTS AND LOCATIONS:
Overall Officials: Julia Seinsche, M.Sc., Principal Investigator — ETH Zürich
Locations (1):
- ETH, Zurich, Switzerland

REFERENCES:
- [Background] Herold F, Hamacher D, Schega L, Muller NG. Thinking While Moving or Moving While Thinking - Concepts of Motor-Cognitive Training for Cognitive Performance Enhancement. Front Aging Neurosci. 2018 Aug 6;10:228. doi: 10.3389/fnagi.2018.00228. eCollection 2018. PMID 30127732
- [Background] Huber SK, Knols RH, Arnet P, de Bruin ED. Motor-cognitive intervention concepts can improve gait in chronic stroke, but their effect on cognitive functions is unclear: A systematic review with meta-analyses. Neurosci Biobehav Rev. 2022 Jan;132:818-837. doi: 10.1016/j.neubiorev.2021.11.013. Epub 2021 Nov 20. PMID 34815131
- [Background] Lauenroth A, Ioannidis AE, Teichmann B. Influence of combined physical and cognitive training on cognition: a systematic review. BMC Geriatr. 2016 Jul 18;16:141. doi: 10.1186/s12877-016-0315-1. PMID 27431673
- [Background] Kraft E. Cognitive function, physical activity, and aging: possible biological links and implications for multimodal interventions. Neuropsychol Dev Cogn B Aging Neuropsychol Cogn. 2012;19(1-2):248-63. doi: 10.1080/13825585.2011.645010. PMID 22313174
- [Background] Tait JL, Duckham RL, Milte CM, Main LC, Daly RM. Influence of Sequential vs. Simultaneous Dual-Task Exercise Training on Cognitive Function in Older Adults. Front Aging Neurosci. 2017 Nov 7;9:368. doi: 10.3389/fnagi.2017.00368. eCollection 2017. PMID 29163146
- [Background] Yang C, Moore A, Mpofu E, Dorstyn D, Li Q, Yin C. Effectiveness of Combined Cognitive and Physical Interventions to Enhance Functioning in Older Adults With Mild Cognitive Impairment: A Systematic Review of Randomized Controlled Trials. Gerontologist. 2020 Nov 23;60(8):633-642. doi: 10.1093/geront/gnz149. PMID 31697831
- [Background] Morat M, Bakker J, Hammes V, Morat T, Giannouli E, Zijlstra W, Donath L. Effects of stepping exergames under stable versus unstable conditions on balance and strength in healthy community-dwelling older adults: A three-armed randomized controlled trial. Exp Gerontol. 2019 Nov;127:110719. doi: 10.1016/j.exger.2019.110719. Epub 2019 Sep 9. PMID 31513877
- [Background] Wuest S, Borghese NA, Pirovano M, Mainetti R, van de Langenberg R, de Bruin ED. Usability and Effects of an Exergame-Based Balance Training Program. Games Health J. 2014 Apr 1;3(2):106-114. doi: 10.1089/g4h.2013.0093. PMID 24804155
- [Background] Swanenburg J, Wild K, Straumann D, de Bruin ED. Exergaming in a Moving Virtual World to Train Vestibular Functions and Gait; a Proof-of-Concept-Study With Older Adults. Front Physiol. 2018 Jul 31;9:988. doi: 10.3389/fphys.2018.00988. eCollection 2018. PMID 30108511
- [Background] Adcock M, Fankhauser M, Post J, Lutz K, Zizlsperger L, Luft AR, Guimaraes V, Schattin A, de Bruin ED. Effects of an In-home Multicomponent Exergame Training on Physical Functions, Cognition, and Brain Volume of Older Adults: A Randomized Controlled Trial. Front Med (Lausanne). 2020 Jan 28;6:321. doi: 10.3389/fmed.2019.00321. eCollection 2019. PMID 32047751
- [Background] Adcock M, Thalmann M, Schattin A, Gennaro F, de Bruin ED. A Pilot Study of an In-Home Multicomponent Exergame Training for Older Adults: Feasibility, Usability and Pre-Post Evaluation. Front Aging Neurosci. 2019 Nov 22;11:304. doi: 10.3389/fnagi.2019.00304. eCollection 2019. PMID 31824295
- [Background] Tillou A, Kelley-Quon L, Burruss S, Morley E, Cryer H, Cohen M, Min L. Long-term postinjury functional recovery: outcomes of geriatric consultation. JAMA Surg. 2014 Jan;149(1):83-9. doi: 10.1001/jamasurg.2013.4244. PMID 24284836
- [Background] Allegue DR, Higgins J, Sweet SN, Archambault PS, Michaud F, Miller W, Tousignant M, Kairy D. Rehabilitation of Upper Extremity by Telerehabilitation Combined With Exergames in Survivors of Chronic Stroke: Preliminary Findings From a Feasibility Clinical Trial. JMIR Rehabil Assist Technol. 2022 Jun 22;9(2):e33745. doi: 10.2196/33745. PMID 35731560
- [Background] Gallou-Guyot M, Nuic D, Mandigout S, Compagnat M, Welter ML, Daviet JC, Perrochon A. Effectiveness of home-based rehabilitation using active video games on quality of life, cognitive and motor functions in people with Parkinson's disease: a systematic review. Disabil Rehabil. 2022 Dec;44(26):8222-8233. doi: 10.1080/09638288.2021.2022780. Epub 2022 Jan 4. PMID 34982599
- [Background] Gandolfi M, Geroin C, Dimitrova E, Boldrini P, Waldner A, Bonadiman S, Picelli A, Regazzo S, Stirbu E, Primon D, Bosello C, Gravina AR, Peron L, Trevisan M, Garcia AC, Menel A, Bloccari L, Vale N, Saltuari L, Tinazzi M, Smania N. Virtual Reality Telerehabilitation for Postural Instability in Parkinson's Disease: A Multicenter, Single-Blind, Randomized, Controlled Trial. Biomed Res Int. 2017;2017:7962826. doi: 10.1155/2017/7962826. Epub 2017 Nov 26. PMID 29333454
- [Background] Md Fadzil NH, Shahar S, Rajikan R, Singh DKA, Mat Ludin AF, Subramaniam P, Ibrahim N, Vanoh D, Mohamad Ali N. A Scoping Review for Usage of Telerehabilitation among Older Adults with Mild Cognitive Impairment or Cognitive Frailty. Int J Environ Res Public Health. 2022 Mar 28;19(7):4000. doi: 10.3390/ijerph19074000. PMID 35409683
- [Background] Rosenberg D, Depp CA, Vahia IV, Reichstadt J, Palmer BW, Kerr J, Norman G, Jeste DV. Exergames for subsyndromal depression in older adults: a pilot study of a novel intervention. Am J Geriatr Psychiatry. 2010 Mar;18(3):221-6. doi: 10.1097/JGP.0b013e3181c534b5. PMID 20173423
- [Background] Tao G, Miller WC, Eng JJ, Lindstrom H, Imam B, Payne M. Self-directed usage of an in-home exergame after a supervised telerehabilitation training program for older adults with lower-limb amputation. Prosthet Orthot Int. 2020 Apr;44(2):52-59. doi: 10.1177/0309364620906272. Epub 2020 Mar 1. PMID 32114933
- [Background] van Diest M, Stegenga J, Wortche HJ, Verkerke GJ, Postema K, Lamoth CJ. Exergames for unsupervised balance training at home: A pilot study in healthy older adults. Gait Posture. 2016 Feb;44:161-7. doi: 10.1016/j.gaitpost.2015.11.019. Epub 2015 Dec 13. PMID 27004651
- [Background] Whitehead AL, Julious SA, Cooper CL, Campbell MJ. Estimating the sample size for a pilot randomised trial to minimise the overall trial sample size for the external pilot and main trial for a continuous outcome variable. Stat Methods Med Res. 2016 Jun;25(3):1057-73. doi: 10.1177/0962280215588241. Epub 2015 Jun 19. PMID 26092476
- [Derived] Seinsche J, de Bruin ED, Saibene E, Rizzo F, Carpinella I, Ferrarin M, Ifanger S, Moza S, Giannouli E. Feasibility and Effectiveness of a Personalized Home-Based Motor-Cognitive Training Program in Community-Dwelling Older Adults: Protocol for a Pragmatic Pilot Randomized Controlled Trial. JMIR Res Protoc. 2023 Nov 9;12:e49377. doi: 10.2196/49377. PMID 37943591